CLINICAL TRIAL: NCT04157166
Title: Evaluation of an Accelerated Body-whole Bone CT Procedure With the CZT "VERITON-CT ™" Camera: a Comparison With the Conventional Full-body 2D Recording Procedure With or Without Complementary Tomoscintigraphy.
Brief Title: Evaluation of an Accelerated Body-whole Bone CT Procedure With the CZT "VERITON-CT ™" Camera
Acronym: OSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: GIE NANCYCLOTEP (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Central HNF
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Bone Metastases
Keywords: Bone scan; solid state gama camera CZT-based detector; hybrid SPECT/CT imaging; bone metastasis

STUDY DESIGN:
Intervention Model Description: a group in which the conventional recording followed by complementary images in planar or TEMP, will be realized in first intention and the procedure of recording of 25 minutes in camera VERITON-CT ™ including the registration whole body 3D coupled to a scanner low dose (CT), will be performed just before and,
  * another group in which these recordings will be made in the reverse order
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 in pair week (Other): In pair week, patients will inclued in group1: the conventional recording followed by complementary images SPECT/CT, will be realized in first intention and the procedure of recording in camera VERITON will be recorderd in second intention
  Interventions: Diagnostic Test: to record a whole body 3D of 25 minutes in camera VERITON-CT ™
- group 2 in odd week (Other): in odd week, patients will inclued in group2: the procedure of recording of 25 minutes in camera VERITON-CT ™, will be realized in first intention and the procedure of conventional recording followed by complementary images SPECT/CT will be recorded in second intention
  Interventions: Diagnostic Test: to record a whole body 3D of 25 minutes in camera VERITON-CT ™

INTERVENTIONS:
Diagnostic Test: to record a whole body 3D of 25 minutes in camera VERITON-CT ™ — The procedure of recording of 25 minutes in camera VERITON-CT ™ including the registration whole body 3D coupled to a scanner low dose (CT) will be added to conventional recording followed by complementary images SPECT/CT

SUMMARY:
The purpose of the OSS study is to evaluate a procedure involving a single full body TEMP / TDM 3D recording with a new semiconductor camera, the VERITON-CT ™ (Spectrum Dynamics Medical). This recording can be done in less than 25 minutes due to an original system of CZT (Cadmium-Zinc-Telluride) detectors allowing to increase the quality of the images and especially, to multiply by a factor 2 to 3 the detection sensitivity. This camera is also equipped with a scanner capable of obtaining a body-to-integer recording with a low level of irradiation (≤ 2 mSv)

DETAILED DESCRIPTION:
Interventional study (RIPH-2), monocentric and randomized in open. All patients routinely referred for bone scans as part of a search for primary or metastatic neoplastic bone lesions (known neoplastic history) will be offered to participate in the study by the doctors of the nuclear medicine department of the CHRU from Nancy.

The capture of tracers used for bone scintigraphy (technetium-99m-labeled bisphosphonates) is highly dependent on bone remodeling, osteoblast activity and tissue perfusion . This is why bone scintigraphy is a sensitive examination, capable of detecting anomalies before their radiological translation . 3-dimensional (3D) recordings called SPECT detect bone metastases with a sensitivity equivalent to that of MRI .

These SPECT are most often produced by hybrid systems, in combination with X-ray scanner (CT) recordings, which makes it possible to correct certain imperfections in the quantification of the measured activities (attenuation, diffusion, partial volume) and also, to complete the characterization of lesions.

Bone diseases, which are often diffuse, frequently require two-dimensional (2D) whole body recordings, but these are unfortunately less informative and less sensitive than 3D recordings. This is why complementary focused SPECT / CT images are recommended for areas that are difficult to explore, especially the pelvis and spine, and when neoplastic lesions are suspected. This registration procedure is long (about 40 minutes), difficult for some patients to support, and does not offer an optimal 3D analysis of the entire skeleton.

ELIGIBILITY:
Inclusion Criteria:

* Patient having read and understood the information document and having signed the consent.
* Patient referred for bone scintigraphy to detect possible metastatic or primary neoplastic lesions (known neoplastic antecedent), or for assessment and / or follow-up of known neoplastic bone lesions
* Patient acceptant de réaliser les 25 minutes d'enregistrement supplémentaire avec la caméra VERITON-CT™.
* Patient being affiliated to a social security scheme

Exclusion Criteria:

* A woman who is pregnant or of childbearing age and without suitable contraceptive means
* No signature of the informed consent form by the patient.
* Unstable medical condition and / or inability to remain still in the supine position during the recordings
* Person with a known allergy to one of the components of the radiotracer (TECHNESCAN HDP).
* Person deprived of liberty by a judicial or administrative decision.
* Major person subject to a legal protection measure (guardianship, curatorship, safeguard of justice).
* Major person unable to express consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2020-01-20 (Estimated); Primary Completion 2021-01-21 (Estimated); Study Completion 2022-01-20 (Estimated)

PRIMARY OUTCOMES:
concordance between the two procedures | half hour
  Concordance between the 2 procedures of the importance of scintigraphic abnormalities evoking a neoplastic process and which will be classified into 3 categories (these categories may correspond to different medical and therapeutic care) : 1) absence of any suspicious focus, 2) 1 or 2 metastases 3) more than 2 metastases

SECONDARY OUTCOMES:
concordance between the two procedures 3D | half hour
  Concordance between the 2 procedures 3D of a same region abnormalities evoking a neoplastic process and which will be classified into 3 categories (these categories may correspond to different medical and therapeutic care) : 1) absence of any suspicious focus, 2) 1 or 2 metastases 3) more than 2 metastases

IPD SHARING:
Plan to Share IPD: No